CLINICAL TRIAL: NCT05420883
Title: Effect of Acupressure and Halogen Light Stimulation on Nonstress Testing and Pregnant Anxiety: A Randomized Controlled Study
Brief Title: The Effect of Acupressure and Halogen Light Stimulation on Nonstress Testing and Pregnant Anxiety
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ondokuz Mayıs University (Other)
Collaborators: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Yasemin Sökmen, Lecturer, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: d5uaw8rc
Record Dates: First submitted 2022-06-05; First posted 2022-06-15 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Acupressure
Keywords: Nonstress test; Anxiety; Halogen light; Acupressure
MeSH Terms: conditions — Anxiety Disorders | interventions — Acupressure

STUDY DESIGN:
Intervention Model Description: Akupresür One minute after the start of the Nonstress test recording, an application will be made to the Zhi yin (BL67) acupuncture point with a depth of 0.1-0.2 cm, on the outer edge of the little toe of both feet, at the nail end point. The application will be applied to both points simultaneously for 2 minutes consecutively and then repeated 2 times with a 3-minute rest period.
  Halojen ışık One minute after the start of the Nonstress Test recording, halogen light stimulation will be given from the mother's abdomen to the fetal head for 10 seconds with a flashlight device worth 1,000,000 candles. The procedure will be repeated on the same spot 10 minutes after the first halogen light stimulation.
  Kontrol No action will be taken against this group.
Who Masked: Participant
Masking Description: Acupressure group One minute after the Nonstress test recording starts, sequential pressure will be applied to the Zhi yin (BL67) acupuncture points simultaneously for 2 minutes. The process will be repeated a second time, with a three-minute rest period. After the 20-minute Nonstress test procedure, the test will be evaluated by the researcher and her anxiety will be determined.
  Halojen ışık group One minute after the start of the Nonstress test recording, halogen light stimulation will be given from the mother's abdomen over the fetal head for 10 seconds and the procedure will be repeated after 10 minutes. After the 20-minute Nonstress test procedure, the test will be evaluated by the researcher and her anxiety will be determined.
  Kontrol Group No application will be made to the control group. After the 20-minute Nonstress test procedure, the test will be evaluated by the researcher and her anxiety will be determined.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Acupressure (Active Comparator): One minute after the start of the Nonstress test recording, an application will be made to the Zhi yin (BL67) acupuncture point with a depth of 0.1-0.2 cm, on the outer edge of the little toe of both feet, at the nail end point. The application will be applied to both points simultaneously for 2 minutes consecutively and then repeated 2 times with a 3-minute rest period.
  Interventions: Other: Halojen ışık; Other: Control
- Halogen light (Active Comparator): One minute after the start of the Nonstress Test recording, halogen light stimulation will be given from the mother's abdomen to the fetal head for 10 seconds with a flashlight device worth 1,000,000 candles. The procedure will be repeated on the same spot 10 minutes after the first halogen light stimulation.
  Interventions: Other: Acupressure; Other: Control
- Control (Active Comparator): No action will be taken against this group.
  Interventions: Other: Acupressure; Other: Halojen ışık

INTERVENTIONS:
Other: Acupressure — One minute after the Nonstress test recording starts, sequential pressure will be applied to the Zhi yin (BL67) acupuncture points simultaneously for 2 minutes. The process will be repeated a second time, with a three-minute rest period. After the 20-minute Nonstress test procedure, the test will be evaluated by the researcher and her anxiety will be determined.
  Arms: Control; Halogen light
Other: Halojen ışık — One minute after the start of the Nonstress test recording, halogen light stimulation will be given from the mother's abdomen over the fetal head for 10 seconds and the procedure will be repeated after 10 minutes. After the 20-minute Nonstress test procedure, the test will be evaluated by the researcher and her anxiety will be determined.
  Arms: Acupressure; Control
Other: Control — No application will be made to the control group. After the 20-minute Nonstress test procedure, the test will be evaluated by the researcher and her anxiety will be determined.
  Arms: Acupressure; Halogen light

SUMMARY:
Fetal death accounts for approximately half of perinatal death. Fetal health should be evaluated in order to identify fetuses at risk of intrauterine death and to prevent perinatal morbidity and mortality. The Nonstress test, which is used to evaluate fetal health, is an important issue as it provides health professionals with information about fetal health. The research was planned as a randomized controlled trial to examine the effect of acupressure and halogen light stimulation on nonstress testing and anxiety of the pregnant woman. The research is planned to be conducted in the nonstress test room of the Obstetrics and Gynecology outpatient clinic of Samsun Training and Research Hospital Gynecology and Childhood Diseases Hospital between May 2021 and June 2023. The sample size of the study was calculated by power analysis (G*Power 3.1.9.2 program was used) and a total of 120 pregnant women were found. In order to increase the analysis power of the research, the number of samples was increased by 20% and it was decided to have at least 144 pregnant women (acupressure group: 48; halogen light group: 48 and control group: 48) for the study. The data of the study will be collected with the Pregnant Identification Form, the Nonstress Test Follow-up Form and the State Anxiety Scale. The data of the study will be evaluated using the SPSS 24 deviation, median and minimum-maximum values will be given. Chi-square test, Student t test, ANOVA test for those with normal distribution, Mann-Whitney U and Kruskal Wallis tests for those who are not.

DETAILED DESCRIPTION:
H01: There was no difference between the nonstress test results of pregnant women who received acupressure and control group pregnant women.

H02: There was no difference between the anxiety levels of the pregnant women who received acupressure and the control group pregnant women.

H03: There is no difference between the nonstress test results of the pregnant women who received halogen light stimulation and the control group pregnant women.

H04: There was no difference between the anxiety levels of pregnant women who received halogen light stimulation and those in the control group.

H05: There is no difference between the nonstress test results of pregnant women who received acupressure and halogen light stimulation.

H06: There was no difference between the anxiety levels of pregnant women who received acupressure and halogen light stimulation.

This study was designed as a randomized controlled experimental study. The research will be carried out between May 2021 and June 2023 in the Nonstress test room in the obstetrics and gynecology outpatient clinic of Samsun Training and Research Hospital Gynecology and Childhood Diseases Hospital affiliated to Samsun Provincial Health Directorate. The universe of the study will be composed of pregnant women who applied to the Nonstress test room for Nonstress test extraction after having a pregnancy follow-up in the obstetrics and gynecology outpatient clinic of Samsun Training and Research Hospital. The sample of the study will be divided into three groups as acupressure group, halogen light group and control group.

The sample size of the study, according to the power analysis (G*Power 3.1.9.2 program was used) using the values of Rahimikian et al.'s (2013) studies, at least 40 people for each group (acupressure group: 40) with 80% power and 5% margin of error. ; halogen light group: 40 and control group: 40), a total of 120 pregnant women were calculated. In order to increase the analysis power of the research, the number of samples was increased by 20% and it was decided to have at least 144 pregnant women (acupressure group: 48; halogen light group: 48 and control group: 48) for the study. A layer will be formed in terms of age, number of pregnancies and gestational week of the pregnant women in the acupressure group, halogen light group and control group, and a homogeneous distribution of the groups will be ensured. Which group the participants will be in will be determined by the full randomization technique on the website www.randomizer.org. After obtaining permission from the ethics committee and the institution that will carry out the study, the pregnant women will go to the institution. Pregnant women who meet the research criteria will be informed about the purpose, content and method of the research, and verbal and written consent will be obtained from those who want to participate. The researcher will meet the pregnant women face to face and fill out the Pregnant Identification Form, the Nonstress Test Follow-up Form and the State Anxiety Scale.

Pregnant Identification Form: This form was developed by the researcher and consists of 20 questions, including 6 questions about the socio-demographic characteristics of pregnant women, 11 questions about their obstetric characteristics, and 3 questions about vital signs.

Nonstress Test Follow-up Form: This form was developed by the researcher and consists of a total of 16 questions, 7 questions that determine the thoughts of pregnant women about Nonstress Test and 9 questions about the findings related to Nonstress Test.

State Anxiety Inventory: The State and Trait Anxiety Inventory was developed by Spielberger et al. in 1970. The Turkish validity and reliability study of the scale was performed by Öner and Le Compte in 1985. The State Anxiety Inventory is a 20-item scale used to determine how an individual feels at a certain moment and under certain conditions. The scale can be administered to individuals over the age of 14 individually or in groups and takes an average of 10 minutes. The scores obtained from the scale theoretically vary between 20 and 80, with a large score indicating a high level of anxiety and a low score indicating a low level of anxiety.

Pre-Practice pre-study will be conducted with ten pregnant women before starting the study to evaluate whether the questions have been understood. As a result of the evaluation, it will be evaluated whether there is a need for editing in the data forms and adjustments will be made. Those included in the preliminary study will not be included in the sample group.

Pregnant women who came for the Nonstress test, met the inclusion criteria and volunteered to participate in the study will be informed about the study and an "Informed Consent Form" will be obtained from those who volunteered to participate in the study. Before starting the Nonstress test, the "Pregnant Identification Form" will be filled in by the researcher by interviewing the pregnant woman face to face. Before the procedure, one fruit juice will be drunk to prevent the difference between the eating times of the pregnant women. Then, the vital signs of the pregnant women will be taken and the fundus height, situs and position will be determined with the Leopold maneuvers by placing the pregnant women in the left lateral recumbent position. According to Leopold maneuver findings, a tocotransducer will be placed at the height of the fundus, and a transducer will be placed at the fetal ridge. Then, a 20-minute NST recording will be started by giving a marker to the pregnant woman's hand.

One minute after the Nonstress test recording starts, the acupressure group will be applied to the Zhi yin (BL67) acupuncture point with a depth of 0.1-0.2 cm, on the outer edge of the little toes of both feet, at the nail end point. The application will be applied to both points consecutively for 2 minutes at the same time and then a 3-minute rest period will be repeated 2 times. Successive pressures will be applied at a frequency that has a calming effect, so that the person is not disturbed or painful. After the nonstress test registration is completed, the State Anxiety Scale will be filled in by the pregnant woman, and the Nonstress Test Follow-up Form will be filled in by the researcher.

The halogen light group will be given halogen light stimulation for 10 seconds from the mother's abdomen to the fetal head one minute after the start of the twenty-minute Nonstress Test recording with a flashlight device (Vector VEC127Y 1 million candle power super sport spotlight with stand) worth 1,000,000 candles. The procedure will be repeated on the same spot 10 minutes after the first halogen light stimulation. After the nonstress test registration is completed, the State Anxiety Scale will be filled in by the pregnant woman, and the Nonstress Test Follow-up Form will be filled in by the researcher.

In the control group, no intervention will be made. The data of the study will be evaluated using the SPSS 24 (PASW Inc., Chicago. IL. USA) program. All data will first be evaluated with Kolmogorov-Smirnov for conformity to normal distribution and then analyzed according to fitness for normal distribution. For descriptive statistics, percentages will be used in general, arithmetic mean±standard deviation for those suitable for normal distribution, median and minimum-maximum values for those that do not fit. Chi-square test, student t test, ANOVA test for those with normal distribution, Mann-Whitney U and Kruskal Wallis tests for those who are not suitable will be used in the analysis of data. Type 1 error level will be taken as 0.05

ELIGIBILITY:
Inclusion Criteria:

* Those between the ages of 18-35,
* Gestational week of 34 and above,
* Single and live pregnancy,
* Number of births ≤3
* Having had Nonstress test at least once before,
* Having regular antenatal follow-up,
* Able to speak and understand Turkish,
* Pregnant women with at least primary school graduates will be included in the study.
* Eating at least two hours before the nonstress test,
* Not using cigarettes, alcohol or drugs at least two hours before the Nonstress test,
* Not doing vigorous activity at least two hours before the Nonstress test,
* Urinating just before the Nonstress test,
* Basal heart rate is 110-160 beats per minute.

Exclusion Criteria:

* Having more than one pregnancy loss,
* Uterine contraction as a result of Nonstress test,
* In any situation that develops acutely during the Nonstress test,
* Those who could not complete the Nonstress test for any reason,
* Psychologically diagnosed (such as depression, schizophrenia)
* Any chronic disease (such as diabetes, hypertension, heart failure)
* Pregnancy complications (such as preeclampsia, gestational diabetes, Rh incompatibility)
* Pregnant with a history of infertility and assisted reproductive techniques,
* A problem defined in the fetus (anomaly, intrauterine growth retardation and cardiovascular disease),
* Pre-pregnancy body mass index calculated as 30 and above,
* Pregnant women who give false or incomplete information will not be included in the study.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 144 (Estimated)
Dates: Start 2022-06-15 (Estimated); Primary Completion 2022-11-15 (Estimated); Study Completion 2022-12-15 (Estimated)

PRIMARY OUTCOMES:
Nonstress test result | "on average 6 months when the study is complete"
  The Nonstress test will be taken for 20 minutes and the result will be evaluated.
Anxiety of the pregnant | "on average 6 months when the study is complete"
  It will be evaluated after the Nonstress test process.

SECONDARY OUTCOMES:
Nonstress test result | An evaluation will be made 20 minutes after the nonstress test process starts.
  The Nonstress test will be taken and the result will be evaluated.
Anxiety of the pregnant | After 20 minutes of Nonstress test
  It will be evaluated after the Nonstress test process.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rahimikian F, Rahiminia T, Modarres M, Mehran A. Comparison of halogen light and vibroacoustic stimulation on nonreactive fetal heart rate pattern. Iran J Nurs Midwifery Res. 2013 Mar;18(2):112-6. PMID 23983739